CLINICAL TRIAL: NCT06414681
Title: An Open Label Pilot Trial of the Combination of Tagraxofusp with Pacritinib in Patients with Intermediate-1 or Higher Myelofibrosis, Who Have Had Prior Therapy with the Approved JAK Inhibitors or in Which Therapy with the Approved JAK Inhibitors is Not Appropriate, Contraindicated or Declined
Brief Title: Combination of Tagraxofusp with Pacritinib in Patients with Intermediate-1 or Higher Myelofibrosis, Who Have Had Prior Therapy with the Approved JAK Inhibitors or in Which Therapy with the Approved JAK Inhibitors is Not Appropriate, Contraindicated or Declined
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Abdulraheem Yacoub, Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00160238
Record Dates: First submitted 2024-02-23; First posted 2024-05-16 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Myelofibrosis，MF
Keywords: Myelofibrosis; MF; JAK 1/2; Tagraxofusp; TAG; Pacritinib; PAC; Tagraxofusp with Pacritinib; Intermediate II Myelofibrosis; Higher Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — tagraxofusp; 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tagrxofusp (IV) in combination with Pacritinib (Oral) (Experimental): Tagraxofusp Patients will receive 12 micrograms/kg of Tagraxofusp (TAG) by IV infusion once daily for 3 consecutive days.
  Pacritinib Pacritinib (PAC) will be given orally, 200 mg twice per day starting at C2D4 and administered continuously (Subsequent cycles start on Day 1 of the Cycle).
  Interventions: Drug: Tagraxofusp; Drug: Pacritinib

INTERVENTIONS:
Drug: Tagraxofusp — Tagraxofusp Patients will receive 12 micrograms/kg of Tagraxofusp (TAG) by IV infusion once daily for 3 consecutive days.
Drug: Pacritinib — Pacritinib Pacritinib (PAC) will be given orally, 200 mg twice per day starting at C2D4 and administered continuously (Subsequent cycles start on Day 1 of the Cycle).

SUMMARY:
The goal of this open-label, single-center, pilot trial is to test the combination of Tagraxofusp (TAG) with Pacritinib (PAC) in patients with intermediate-II or higher myelofibrosis (MF), who have had prior therapy with the approved JAK1/2 inhibitor or in which therapy with the approved JAK1/2 inhibitors is not appropriate, contraindicated or declined by the subjects.

The Primary Objective is to:

1. Characterized efficacy of the combination of Tagraxofusp and Pacritinib.

The Secondary Objective is to:

1. characterize the safety profile of the combination Tagraxofusp and Pacritinib.

2, Characterize the feasibility of the combination Tagraxofusp and Pacritinib. 3. Characterize hematologic improvement with the combination Tagraxofusp and Pacritinib.

4. Evaluate and compare the effect of Tagraxofusp and Pacritinib on participant reports of MF symptoms.

Exploratory:

Pharmacokinetic (PK) testing of Tagraxofusp and Pacritinib to assess clinical predictors of response.

Next Generation Sequencing (NGS) Testing to define the number and the allele burden of pathological mutations, as well as the changes over the course of therapy, both in regard to progression and response.

Blood will be collected and stored at KU BRCF for future study related PK analysis

DETAILED DESCRIPTION:
A combination of these agent provides rational scientific merit and compatible mechanisms of action by targeting myelofibrosis stem cells and BM environment, in combination with effective JAK2 and IRAK1 inhibition resulting in improvement in MPN related symptoms and splenomegaly without overlapping toxicities. Both agents have been studied in mildly depleted bone marrow phenotypes showing safety and hematological improvements

ELIGIBILITY:
Inclusion Criteria:

1. Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent.
2. The participant or LAR has signed informed consent prior to initiation of any study-specific procedures or treatment.
3. The patient is able to adhere to the study visit schedule and other protocol requirements.
4. Males and females age ≥ 18 years.
5. ECOG Performance Status 0 - 2 (Appendix A).
6. Life expectancy of > 6 months.
7. Patient meets the 2016 WHO diagnostic criteria for MF and has an IPSS/DIPSS/DIPSS-plus intermediate-II or higher-risk disease.
8. Patients who have indications for therapy per investigator or patient's choice, such as Splenomegaly, >5 CM BCM or mTSS ≥ 8 or mTSS Itching, night sweats, or bone pain ≥ 5 or Significant cytopenias including Hgb <10 g/dl, Platelet count less than 75 k/UL
9. Patients treated with a JAK inhibitor for >3 months and:

   had inadequate response to treatment, i.e., < 10% reduction of spleen by imaging, or less than 25% reduction by spleen length on physical exam or lack of control of MF symptoms that is not satisfactory to the patient. NOTE: Participants who had contraindication to therapy with the approved JAK inhibitor including subject's refusal of therapy are eligible.
10. A least 4 weeks have elapsed between the last dose of any MF-directed drug treatments, including hydroxyurea (HU), Interferon or glucocorticosteroids. NOTE: If patient is on a stable dose of glucocorticosteroids for another indication, they will be allowed into this study, AND patients on a stable dose of erythropoiesis-stimulating agents (ESA) are allowed on the study.
11. Patient is not eligible for an immediate allo-SCT.
12. Adequate baseline organ, cardiac, and renal function as defined by:

    LVEF ≥ 50% by ECHO within 6 months of study treatment initiation No clinically significant abnormalities on a 12-lead ECG, and no QTcF ≥ 480 msec Serum creatinine ≤ 1.5 mg/dL Serum albumin ≥ 3.2 g/dL (Note: albumin infusions are not permitted to enable eligibility) INR and PTT ≤ 1.5x ULN Albumin Supplementation Prior to the first dose, participant must have serum albumin ≥ to 3.2 g/dL.

    Note- for any participants with serum albumin ≤ to 4.0 g/dL, it will be advisable but up to physician's discretion to administer 25g increments of albumin infusion before the first dose.

    Total bilirubin ≤ 4x ULN AST and ALT ≤ 5 x ULN ANC ≥ 0.5 x 109/L PT or INR and PTT < = 1.5 x ULN
13. If the patient is a woman of child-bearing potential (WOCBP), they should have a negative serum pregnancy test no more than 7 days prior to start of treatment.

    (Note: WOCBP include any female who has experienced menarche and who has not undergone successful sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea ≥ 12 consecutive months; or women on hormone replacement therapy with documented serum follicle stimulating hormone level ≥ 35 mIU/mL).
14. Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence or to use the forms of contraception listed in Child-Bearing Potential/Pregnancy section for the duration of study participation and for 3 months following completion of therapy.

Exclusion Criteria:

1. Simultaneously enrolled in any therapeutic clinical trial
2. Current or anticipating use of other anti-neoplastic or investigational agents while participating in this study.
3. The patient has received treatment with chemotherapy, wide-field radiation, or biologic therapy within 14 days of study entry.
4. The patient has received treatment with another investigational agent within 14 days of study entry.
5. Diagnosed with a psychiatric illness or is in a social situation that would limit compliance with study requirements.
6. Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, disseminated intravascular coagulation.
7. Any condition or other contraindication to therapy as deemed by the principal investigator to place the subject at an unacceptably high risk for toxicities.
8. Is pregnant or breastfeeding.
9. Has a known allergic reaction to any excipient contained in the study drug formulation.
10. Active Grade 3 (per the NCI CTCAE, Version 5.0) or higher viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study treatment.
11. Prior therapy with Tagraxofusp or Pacritinib.
12. Presence of peripheral blood or bone marrow blast count > 10%
13. Active Graft versus Host Disease (GVHD)
14. For patients who have previously had Stem Cell Therapy (SCT) - The patient is receiving immunosuppressive therapy.

    EXCEPTION: low-dose prednisone (≤10 mg/day) - for treatment or prophylaxis of graft-versus-host disease (GVHD). If the patient has been on immunosuppressive treatment or prophylaxis for GVHD, the treatment(s) must have been discontinued at least 14 days prior to study treatment and there must be no evidence of Grade ≥ 2 GVHD.
15. Other uncontrolled active malignancy as determined by the principal investigator
16. The patient has an active malignancy and/or cancer history that may confound the assessment of the study endpoints. Patients with a past cancer history (within 2 years of entry) with substantial potential for recurrence and/or ongoing active malignancy must be discussed with the Sponsor before study entry. Patients with the following neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ, cervical intraepithelial neoplasia, organ-confined prostate cancer with no evidence of progressive disease.
17. The patient has clinically significant cardiovascular disease (e.g. uncontrolled or any New York Heart Association Class 2 or greater congestive heart failure, uncontrolled angina, history of myocardial infarction, unstable angina or stroke within 6 months prior to study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication).
18. Any gastrointestinal or metabolic condition that could interfere with absorption of oral medication.
19. Prior therapy with Pacritinib (PAC) or Tagraxofusp (TAG).
20. The patient has persistent clinically significant toxicities Grade ≥ 2 from previous therapies, including cytotoxic chemotherapy, targeted therapies, biological therapies, or immunotherapies, not readily controlled by supportive measures (excluding alopecia, nausea, and fatigue).
21. The patient has uncontrolled, clinically significant pulmonary disease (e.g. chronic obstructive pulmonary disease, pulmonary hypertension) that in the opinion of the Investigator would put the patient at significant risk for pulmonary complications during the study.
22. The patient has known active or suspected central nervous system (CNS) disease. If suspected, CNS disease should be ruled out with relevant imaging and/or examination of cerebrospinal fluid.
23. Current systemic treatment with strong or moderate CYP3A4 inhibitor or P450 inducer.

    EXCEPTION: Patients who discontinue this treatment by Day 14 before start of treatment (Day -14) or 5 half-lives, whichever is shorter.
24. Use of full-dose anticoagulation and use of anti-platelet therapy other than aspirin 81mg daily within 14 days prior to D1.
25. Recent unprovoked bleeding of grade ≥ 2 within the last 3 months prior to Day 1.
26. Active uncontrolled diarrhea or inflammatory bowel disease (IBD)
27. Known sero-positivity for Hepatitis A (HAV), Hepatitis B (HBV), Hepatitis C (HCV), Human Immunodeficiency Virus (HIV)
28. Patients with history of clinically significant bleeding or on anticoagulants
29. Patients with moderate (Child-Pugh B ) and severe (Child -Pugh C) hepatic impairment will not be enrolled in the study.
30. Patients with eGFR < 30 mL/min will not be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-28 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Spleen volume reduction by MRI or CT imaging, achieving ≥ 35% reduction in spleen volume imaging from baseline to week 24. | Baseline to up to 24 weeks
  MRI of abdomen will be performed WITHOUT contrast. If MRI is contraindicated - CT scan will be allowed (IV contrast will be used unless contraindicated). The same type of Imaging used at screening must continue to be used throughout the study.
Change from baseline in the Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score Version 2.0 (MPN-SAF TSS 2.0) to week 24. | Baseline to up to 24 weeks
  Improvement in symptoms: >/= 50% reduction in Modified Total Symptom Score (mTSS) from baseline to week 24 as measured by the Myeloproliferative Neoplasms Symptom Assessment Form Total Symptom Score Version 2.0 (MPN-SAF TSS 2.0). The MPN Symptom Assessment Form) includes the assessment of symptoms that are relevant to myelofibrosis. MPN-SAF was simplified to a concise and abbreviated tool called the MPN-SAF Total Symptom Score (MPN-SAF TSS), that is used for the assessment of the 10 most relevant symptoms in subjects with MPN (fatigue, concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss, and fever) in both clinical practice and clinical trial settings. The symptom severity is rated by subjects on a scale of 1 to10 MPN-SAF-TSS: a total score will be calculated by the addition of every individual symptom score. The change from baseline will be statically measured and reported.

SECONDARY OUTCOMES:
Number of participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 from baseline to End of Safety Follow-up (30 days after end of treatment). | Baseline to End of Safety follow up to End of Treatment (up to 1 year)
  Number of participants with treatment related adverse events a assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Change from baseline in Anemia (hemoglobin GM/DL, iron ug/DL, and hematocrit %) improvement within or at 1 year | Baseline, Week 24 and End of Treatment (up to 1 year)
  From Baseline to best response within 1 year
Patient's Global Impression (perception) of Change | Every cycle (each cycle is 28 days) day 1 starting at Cycle 2 to End of Treatment (up to 1 year)
Improvement in Quality of Life based on Patient Impression of Global Change (PGIC). A PGIC score of 2 for "much improved" or a score of 1 for "very much improved." | Baseline to up to 24 weeks
  Based on the proportion of patients who report "much improved" or "very much improved" symptoms at Week 24 based on the Patient Impression of Global Change (PGIC). A PGIC score of 2 for "much improved" or a score of 1 for "very much improved."
  The PGIC uses a score between 1 and 7 (1 being "very much improved" to 7 being "very much worse)."
Change from baseline in platelet count in K/UL within 1 year | Baseline, up to 24 weeks and End of Treatment (up to 1 year)
  From Baseline to best response within 1 year
Change from baseline in Anemia (iron ug/DL) | Baseline, Week 24 and End of Treatment (up to 1 year)
  From Baseline to best response within 1 year
Change from baseline in Anemia (hematocrit %) | Baseline, Week 24 and End of Treatment (up to 1 year)
  From Baseline to best response within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Abdulraheem Yacoub, Doctor of Medicine, Principal Investigator — University of Kansas Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Korinek J. [Serum hemopexin values of patients with various diseases and reflection on the probable role of hemopexin in the organizm] (Cze) FLECTION ON THE PROBABLE ROLE OF HEMOPEXIN IN THE ORGANISM]. Cas Lek Cesk. 1969 Jul 18;108(31):919-23. No abstract available. Czech. PMID 4979167
- [Background] Jordan CT, Guzman ML, Noble M. Cancer stem cells. N Engl J Med. 2006 Sep 21;355(12):1253-61. doi: 10.1056/NEJMra061808. No abstract available. PMID 16990388
- [Background] Hurst H, Bolton J. Assessing the clinical significance of change scores recorded on subjective outcome measures. J Manipulative Physiol Ther. 2004 Jan;27(1):26-35. doi: 10.1016/j.jmpt.2003.11.003. PMID 14739871
- [Background] Tefferi A. Challenges facing JAK inhibitor therapy for myeloproliferative neoplasms. N Engl J Med. 2012 Mar 1;366(9):844-6. doi: 10.1056/NEJMe1115119. No abstract available. PMID 22375977
- [Background] Tefferi A. Primary myelofibrosis: 2013 update on diagnosis, risk-stratification, and management. Am J Hematol. 2013 Feb;88(2):141-50. doi: 10.1002/ajh.23384. PMID 23349007
- [Background] Barosi G, Tefferi A, Besses C, Birgegard G, Cervantes F, Finazzi G, Gisslinger H, Griesshammer M, Harrison C, Hehlmann R, Hermouet S, Kiladjian JJ, Kroger N, Mesa R, Mc Mullin MF, Pardanani A, Passamonti F, Samuelsson J, Vannucchi AM, Reiter A, Silver RT, Verstovsek S, Tognoni G, Barbui T. Clinical end points for drug treatment trials in BCR-ABL1-negative classic myeloproliferative neoplasms: consensus statements from European LeukemiaNET (ELN) and Internation Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT). Leukemia. 2015 Jan;29(1):20-6. doi: 10.1038/leu.2014.250. Epub 2014 Aug 25. PMID 25151955
- [Background] Harrison C, Kiladjian JJ, Al-Ali HK, Gisslinger H, Waltzman R, Stalbovskaya V, McQuitty M, Hunter DS, Levy R, Knoops L, Cervantes F, Vannucchi AM, Barbui T, Barosi G. JAK inhibition with ruxolitinib versus best available therapy for myelofibrosis. N Engl J Med. 2012 Mar 1;366(9):787-98. doi: 10.1056/NEJMoa1110556. PMID 22375970
- [Background] Harrison CN, Mesa RA, Kiladjian JJ, Al-Ali HK, Gisslinger H, Knoops L, Squier M, Sirulnik A, Mendelson E, Zhou X, Copley-Merriman C, Hunter DS, Levy RS, Cervantes F, Passamonti F, Barbui T, Barosi G, Vannucchi AM. Health-related quality of life and symptoms in patients with myelofibrosis treated with ruxolitinib versus best available therapy. Br J Haematol. 2013 Jul;162(2):229-39. doi: 10.1111/bjh.12375. Epub 2013 May 14. PMID 23672349
- [Background] Verstovsek S, Mesa RA, Gotlib J, Levy RS, Gupta V, DiPersio JF, Catalano JV, Deininger M, Miller C, Silver RT, Talpaz M, Winton EF, Harvey JH Jr, Arcasoy MO, Hexner E, Lyons RM, Paquette R, Raza A, Vaddi K, Erickson-Viitanen S, Koumenis IL, Sun W, Sandor V, Kantarjian HM. A double-blind, placebo-controlled trial of ruxolitinib for myelofibrosis. N Engl J Med. 2012 Mar 1;366(9):799-807. doi: 10.1056/NEJMoa1110557. PMID 22375971
- [Background] Mughal TI, Cross NC, Padron E, Tiu RV, Savona M, Malcovati L, Tibes R, Komrokji RS, Kiladjian JJ, Garcia-Manero G, Orazi A, Mesa R, Maciejewski JP, Fenaux P, Itzykson R, Mufti G, Solary E, List AF. An International MDS/MPN Working Group's perspective and recommendations on molecular pathogenesis, diagnosis and clinical characterization of myelodysplastic/myeloproliferative neoplasms. Haematologica. 2015 Sep;100(9):1117-30. doi: 10.3324/haematol.2014.114660. PMID 26341525
- [Background] Barbui T, Tefferi A, Vannucchi AM, Passamonti F, Silver RT, Hoffman R, Verstovsek S, Mesa R, Kiladjian JJ, Hehlmann R, Reiter A, Cervantes F, Harrison C, Mc Mullin MF, Hasselbalch HC, Koschmieder S, Marchetti M, Bacigalupo A, Finazzi G, Kroeger N, Griesshammer M, Birgegard G, Barosi G. Philadelphia chromosome-negative classical myeloproliferative neoplasms: revised management recommendations from European LeukemiaNet. Leukemia. 2018 May;32(5):1057-1069. doi: 10.1038/s41375-018-0077-1. Epub 2018 Feb 27. PMID 29515238
- [Background] Prager BC, Xie Q, Bao S, Rich JN. Cancer Stem Cells: The Architects of the Tumor Ecosystem. Cell Stem Cell. 2019 Jan 3;24(1):41-53. doi: 10.1016/j.stem.2018.12.009. PMID 30609398
- [Background] Desai A, Yan Y, Gerson SL. Concise Reviews: Cancer Stem Cell Targeted Therapies: Toward Clinical Success. Stem Cells Transl Med. 2019 Jan;8(1):75-81. doi: 10.1002/sctm.18-0123. Epub 2018 Oct 17. PMID 30328686
- [Background] Yan B, Chen Q, Shimada K, Tang M, Li H, Gurumurthy A, Khoury JD, Xu B, Huang S, Qiu Y. Histone deacetylase inhibitor targets CD123/CD47-positive cells and reverse chemoresistance phenotype in acute myeloid leukemia. Leukemia. 2019 Apr;33(4):931-944. doi: 10.1038/s41375-018-0279-6. Epub 2018 Oct 5. PMID 30291336
- [Background] Arai N, Homma M, Abe M, Baba Y, Murai S, Watanuki M, Kawaguchi Y, Fujiwara S, Kabasawa N, Tsukamoto H, Uto Y, Ariizumi H, Yanagisawa K, Hattori N, Saito B, Shiozawa E, Harada H, Yamochi-Onizuka T, Nakamaki T, Takimoto M. Impact of CD123 expression, analyzed by immunohistochemistry, on clinical outcomes in patients with acute myeloid leukemia. Int J Hematol. 2019 May;109(5):539-544. doi: 10.1007/s12185-019-02616-y. Epub 2019 Mar 7. PMID 30847774
- [Background] Stevens BM, Zhang W, Pollyea DA, Winters A, Gutman J, Smith C, Budde E, Forman SJ, Jordan CT, Purev E. CD123 CAR T cells for the treatment of myelodysplastic syndrome. Exp Hematol. 2019 Jun;74:52-63.e3. doi: 10.1016/j.exphem.2019.05.002. Epub 2019 May 25. PMID 31136781
- [Background] Jordan CT, Upchurch D, Szilvassy SJ, Guzman ML, Howard DS, Pettigrew AL, Meyerrose T, Rossi R, Grimes B, Rizzieri DA, Luger SM, Phillips GL. The interleukin-3 receptor alpha chain is a unique marker for human acute myelogenous leukemia stem cells. Leukemia. 2000 Oct;14(10):1777-84. doi: 10.1038/sj.leu.2401903. PMID 11021753
- [Background] Tehranchi R, Woll PS, Anderson K, Buza-Vidas N, Mizukami T, Mead AJ, Astrand-Grundstrom I, Strombeck B, Horvat A, Ferry H, Dhanda RS, Hast R, Ryden T, Vyas P, Gohring G, Schlegelberger B, Johansson B, Hellstrom-Lindberg E, List A, Nilsson L, Jacobsen SE. Persistent malignant stem cells in del(5q) myelodysplasia in remission. N Engl J Med. 2010 Sep 9;363(11):1025-37. doi: 10.1056/NEJMoa0912228. PMID 20825315
- [Background] Aldinucci D, Olivo K, Lorenzon D, Poletto D, Gloghini A, Carbone A, Pinto A. The role of interleukin-3 in classical Hodgkin's disease. Leuk Lymphoma. 2005 Mar;46(3):303-11. doi: 10.1080/10428190400013712. PMID 15621820
- [Background] Munoz L, Nomdedeu JF, Lopez O, Carnicer MJ, Bellido M, Aventin A, Brunet S, Sierra J. Interleukin-3 receptor alpha chain (CD123) is widely expressed in hematologic malignancies. Haematologica. 2001 Dec;86(12):1261-9. PMID 11726317
- [Background] Aldinucci D, Poletto D, Gloghini A, Nanni P, Degan M, Perin T, Ceolin P, Rossi FM, Gattei V, Carbone A, Pinto A. Expression of functional interleukin-3 receptors on Hodgkin and Reed-Sternberg cells. Am J Pathol. 2002 Feb;160(2):585-96. doi: 10.1016/S0002-9440(10)64878-X. PMID 11839579
- [Background] Black JH, McCubrey JA, Willingham MC, Ramage J, Hogge DE, Frankel AE. Diphtheria toxin-interleukin-3 fusion protein (DT(388)IL3) prolongs disease-free survival of leukemic immunocompromised mice. Leukemia. 2003 Jan;17(1):155-9. doi: 10.1038/sj.leu.2402744. PMID 12529673
- [Background] Frolova O, Frankel AE, Korchin B, et al. IL3R-Directed Agents, SL-401 and SL-501, Inhibit the Growth of Leukemia Stem cells in CML. Blood (ASH Meeting Abstracts) 2010 116: Abstract 3403
- [Background] Florian S, Sonneck K, Hauswirth AW, Krauth MT, Schernthaner GH, Sperr WR, Valent P. Detection of molecular targets on the surface of CD34+/CD38-- stem cells in various myeloid malignancies. Leuk Lymphoma. 2006 Feb;47(2):207-22. doi: 10.1080/10428190500272507. PMID 16321850
- [Background] Lhermitte L, de Labarthe A, Dupret C, Lapillonne H, Millien C, Landman-Parker J, Hermine O, Baruchel A, Sigaux F, Macintyre E, Asnafi V. Most immature T-ALLs express Ra-IL3 (CD123): possible target for DT-IL3 therapy. Leukemia. 2006 Oct;20(10):1908-10. doi: 10.1038/sj.leu.2404349. Epub 2006 Aug 10. No abstract available. PMID 16900212
- [Background] Vergez F, Green AS, Tamburini J, Sarry JE, Gaillard B, Cornillet-Lefebvre P, Pannetier M, Neyret A, Chapuis N, Ifrah N, Dreyfus F, Manenti S, Demur C, Delabesse E, Lacombe C, Mayeux P, Bouscary D, Recher C, Bardet V. High levels of CD34+CD38low/-CD123+ blasts are predictive of an adverse outcome in acute myeloid leukemia: a Groupe Ouest-Est des Leucemies Aigues et Maladies du Sang (GOELAMS) study. Haematologica. 2011 Dec;96(12):1792-8. doi: 10.3324/haematol.2011.047894. Epub 2011 Sep 20. PMID 21933861
- [Background] van Rhenen A, Feller N, Kelder A, Westra AH, Rombouts E, Zweegman S, van der Pol MA, Waisfisz Q, Ossenkoppele GJ, Schuurhuis GJ. High stem cell frequency in acute myeloid leukemia at diagnosis predicts high minimal residual disease and poor survival. Clin Cancer Res. 2005 Sep 15;11(18):6520-7. doi: 10.1158/1078-0432.CCR-05-0468. PMID 16166428
- [Background] Lucas N, Duchmann M, Rameau P, Noel F, Michea P, Saada V, Kosmider O, Pierron G, Fernandez-Zapico ME, Howard MT, King RL, Niyongere S, Diop MK, Fenaux P, Itzykson R, Willekens C, Ribrag V, Fontenay M, Padron E, Soumelis V, Droin N, Patnaik MM, Solary E. Biology and prognostic impact of clonal plasmacytoid dendritic cells in chronic myelomonocytic leukemia. Leukemia. 2019 Oct;33(10):2466-2480. doi: 10.1038/s41375-019-0447-3. Epub 2019 Mar 20. PMID 30894665
- [Background] Rapoport AP, Luhowskyj S, Doshi P, DiPersio JF. Mutational analysis of the alpha subunit of the human interleukin-3 receptor. Blood. 1996 Jan 1;87(1):112-22. PMID 8547632
- [Background] Ratts R, Trujillo C, Bharti A, vanderSpek J, Harrison R, Murphy JR. A conserved motif in transmembrane helix 1 of diphtheria toxin mediates catalytic domain delivery to the cytosol. Proc Natl Acad Sci U S A. 2005 Oct 25;102(43):15635-40. doi: 10.1073/pnas.0504937102. Epub 2005 Oct 17. PMID 16230620
- [Background] Kochi SK, Collier RJ. DNA fragmentation and cytolysis in U937 cells treated with diphtheria toxin or other inhibitors of protein synthesis. Exp Cell Res. 1993 Sep;208(1):296-302. doi: 10.1006/excr.1993.1249. PMID 8359223
- [Background] Pemmaraju N, Lane AA, Sweet KL, Stein AS, Vasu S, Blum W, Rizzieri DA, Wang ES, Duvic M, Sloan JM, Spence S, Shemesh S, Brooks CL, Balser J, Bergstein I, Lancet JE, Kantarjian HM, Konopleva M. Tagraxofusp in Blastic Plasmacytoid Dendritic-Cell Neoplasm. N Engl J Med. 2019 Apr 25;380(17):1628-1637. doi: 10.1056/NEJMoa1815105. PMID 31018069
- [Background] Mesa RA, Vannucchi AM, Mead A, Egyed M, Szoke A, Suvorov A, Jakucs J, Perkins A, Prasad R, Mayer J, Demeter J, Ganly P, Singer JW, Zhou H, Dean JP, Te Boekhorst PA, Nangalia J, Kiladjian JJ, Harrison CN. Pacritinib versus best available therapy for the treatment of myelofibrosis irrespective of baseline cytopenias (PERSIST-1): an international, randomised, phase 3 trial. Lancet Haematol. 2017 May;4(5):e225-e236. doi: 10.1016/S2352-3026(17)30027-3. Epub 2017 Mar 20. PMID 28336242
- [Background] Mascarenhas J, Hoffman R, Talpaz M, Gerds AT, Stein B, Gupta V, Szoke A, Drummond M, Pristupa A, Granston T, Daly R, Al-Fayoumi S, Callahan JA, Singer JW, Gotlib J, Jamieson C, Harrison C, Mesa R, Verstovsek S. Pacritinib vs Best Available Therapy, Including Ruxolitinib, in Patients With Myelofibrosis: A Randomized Clinical Trial. JAMA Oncol. 2018 May 1;4(5):652-659. doi: 10.1001/jamaoncol.2017.5818. PMID 29522138
- [Background] Stemline Therapeutics, Inc. ELZONRIS (Tagraxofusp-erzs) Investigator's Brochure Version 6.0 dated 04-20-2021
- [Background] CTI Biopharma Corp. Pacritinib (SB1518) Investigator Brochure (IND 78,4806) Version 13 dated 02-27-2020
- [Background] Stemline Therapeutics. Tagraxofusp Protocol Guidance for the Investigator. Version 2.0 dated 09-29-2021. Provided by Stemline Therapeutics
- [Background] CTI Biopharma Corp. VONJO (Pacritinib) Package Insert dated 02-2022
- [Background] Stemline Therapeutics, Inc. Protocol Number STML-401-0314 Amendment 8 dated 05-05-2020. Tagraxofusp (SL-401) in Patients with Chronic Myelomonocytic Leukemia (CMML) or Myelofibrosis (MF)
- See also: U.S Food and Drug Administration - News and Events for Human Drugs. FDA approves drug for adults with rare form of bone marrow disorder — https://www.fda.gov/drugs/news-events-human-drugs/fda-approves-drug-adults-rare-form-bone-marrow-disorder
- See also: Pacritinib Granted Accelerated Approval for Use in Myelofibrosis With Severe Thrombocytopenia — https://www.cancernetwork.com/view/Pacritinib-granted-accelerated-approval-for-use-in-myelofibrosis-with-severe-thrombocytopenia
- See also: U.S. Food & Drug Administration. For Healthcare Professionals | FDA's Examples of Drugs that Interact with CYP Enzymes and Transporter Systems — https://www.fda.gov/drugs/drug-interactions-labeling/healthcare-professionals-fdas-examples-drugs-interact-cyp-enzymes-and-transporter-systems